CLINICAL TRIAL: NCT04093427
Title: Einfluss Einer Inversen Druckrampe Bei Der Langzeit-Therapie Mit Nicht-invasiver Ventilation Auf Dyspnoe am Morgen Nach Therapie-Ende. Influence of an Inverse Pressure Ramp in the Long-term Therapy Mit Non-invasive Ventilation on Dyspnea in the Morning After Therapy.
Brief Title: Influence of an Inverse Pressure Ramp in Long-term Non-invasive Ventilation on Dyspnea in the Morning After Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment in a timely manner
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Löwenstein Medical Technology GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WI_19-090_softSTOPP
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Noninvasive Ventilation; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- softSTOPP active (Active Comparator)
  Interventions: Other: softSTOPP
- softSTOPP inactive (No Intervention)

INTERVENTIONS:
Other: softSTOPP — Non-invasive ventilation device setting in prismaVENT 30 device enabling an inverse pressure ramp after therapy end
  Arms: softSTOPP active

SUMMARY:
Patients being treated with non-invasive home mechanical ventilation (NIV) may experience morning dyspnea after each night of NIV use, when the therapy is abruptly ended. This study aims to show that dyspnea intensity can be significantly reduced by a gentle NIV therapy end, delivered by a continuously decreasing pressure level (inverse pressure ramp) after therapy end in the morning, a feature called softSTOPP, which can configured in prismaVENT NIV devices. This could also improve therapy adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of a chronic obstructive pulmonary disease (COPD) with chronic hypercapnic insufficiency
* Therapy with prismaVENT 30, firmware V 3.3 or higher, mode S/T, stable device settings at the time of inclusion without need to adapt ventilation parameters
* May have co-existing obstructive sleep apnea syndrome
* Subjective dyspnea ≥3 (Borg scale) after end of ventilation therapy in the morning
* Written informed consent for study participation including data protection

Exclusion Criteria:

* Missing written informed consent for study participation including data protection
* Contraindication for positive airway pressure therapy
* Use of the softSTOPP feature before study inclusion
* Participation in another study, which influences NIV therapy by defining device settings or titration
* Concomitant oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change of dyspnea level from baseline to 12 weeks | 12 weeks
  Delta value of morning dyspnea from baseline to 12 weeks as measured by the Borg Scale. The Borg Scale ranges from 0 (no perceived dyspnea at all) to 10 (maximum perceived dyspnea).

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Krankenhaus Bethanien
Locations (1):
- Krankenhaus Bethanien, Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No